CLINICAL TRIAL: NCT06831318
Title: Community Health Worker-Led Hospital-to-Community Transition Support for Persons Living With Dementia and Their Caregivers
Brief Title: Community Health Worker-Led Transition Support for Persons Living With Dementia and Caregivers
Acronym: CEDART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004286
Record Dates: First submitted 2025-02-04; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Cognitive Impairment; Dementia; Memory Deficits
Keywords: caregiver; care transition; community health worker; dementia; cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Memory Disorders | interventions — Community Health Workers

STUDY DESIGN:
Intervention Model Description: This study is a single-site, single-arm feasibility study with between 40 and 80 hospitalized dyads receiving the CHW-led Care Transition Intervention to obtain preliminary data on the intervention's acceptability, feasibility, and potential efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHW intervention group (Experimental): dementia patient and caregiver dyad
  Interventions: Behavioral: Community Health Worker (CHW) Guided Support

INTERVENTIONS:
Behavioral: Community Health Worker (CHW) Guided Support — The CHW conducts a family assessment, which identifies caregiving stressors, social support, and needs as related to social determinants of health, dementia education, care navigation, caregiver health and burden. Closer to discharge, dyads receive an individualized dementia caregiving toolkit including the post-discharge care planning checklist, tracking sheets for patient medications, tests, and procedures, and info on local resources. All meetings will be done in person, telephone, or zoom.
  Within one week of discharge, the CHW meets the dyad via phone or Zoom to review their goals and to identify any additional needs for coaching, education, or navigation support. In the first month after discharge, the CHW provides weekly or bi-weekly check-ins. For the next two months, the CHW provides about four additional bi-weekly check-in sessions. Each check-in session will last approximately 30-45 minutes. The exact number of meetings will be determined by need and caregiver availability

SUMMARY:
The main purpose of this intervention study is to test if the community health worker (CHW)-led care transition support intervention is feasible and acceptable to the persons living with dementia (PLWD)'s caregivers, and other healthcare providers.

Main hypotheses of the study are:

1. the CHW interventionist will adhere to the intervention protocol with the score of 80% or higher on the intervention fidelity checklist throughout the intervention delivery period;
2. caregiver participants in the intervention group will rate the intervention, and the CHW interventionist to be helpful and satisfactory at the end of the intervention;
3. intervention feasibility (as measured by intervention completion rate, i.e., number of participants completing the telephone sessions with the CHW coach, and participant assessment completion rate, i.e., number of participants completing each study assessment at baseline, 6, 12 weeks) will be at equal to or higher than 80%; and
4. intervention participants - patient and caregiver - outcomes will improve at post-discharge Week 12 follow up from baseline and Week 6.

DETAILED DESCRIPTION:
This study is a single-site, single-arm feasibility study with hospitalized person living with dementia (PLWD) and their family caregiver dyads receiving the community health worker (CHW)-led Care Transition Intervention to obtain preliminary data on the intervention's acceptability, feasibility, and potential efficacy. In addition to evaluation PLWD and caregiver outcomes, multiple stakeholders from two hospitals (Dell Seton Medical Center and Ascension Seton Medical Center Austin) will be interviewed focusing on intervention relevance for healthcare system and provider stakeholder priorities and feasibility and acceptability of integration into everyday workflows. Mixed methods (individual interviews, chart reviews) study will be conducted to gather views of various stakeholders at two hospital sites including PLWD and family caregivers, frontline providers and care staff, administrators, and information technology staff.

Of the two hospitals, Dell Seton Medical Center and Ascension Seton Medical Center Austin, Dell Seton Medical Center (DSMC) will be the main study site where the intervention and recruitment of dyads will take place. At Ascension Seton Medical Center Austin (ASMCA), staff will be interviewed to assess the feasibility and acceptability of the intervention to determine if future implementation at ASMCA is possible.

PLWD and caregiver target enrollment for this study is 80 English- or Spanish-speaking family caregivers and 80 of their care recipients who meet the eligibility criteria. The intervention will be led by a bilingual (English and Spanish speaking) CHW who is trained in the intervention.

The intervention process starts with the family assessment by the CHW, which identifies primary and secondary caregiving stressors, resources and social support availability, and needs for support as related to social determinants of health, dementia education, care navigation, caregiver health and burden. Closer to discharge, the CHW will again make contact with the family caregiver to review the post-discharge care plan and to help the family caregiver develop a plan for post-discharge care. Dyads will receive a curated individualized dementia caregiving toolkit. All meetings with the caregiver during patient's hospitalization will be done in person, via telephone or via zoom, whichever the caregiver prefers. Within the first week of discharge, the CHW will meet via telephone or Zoom with the dyad to review the goals, additional support needs such as care navigation, access to social services, and any other concerns. During the first month after discharge, the CHW will continue to provide weekly or bi-weekly telephone/zoom check-ins as needed for coaching, focused dementia and caregiving education, or navigation support, and provide approximately four additional bi-weekly check-in sessions with the caregiver for the following two months. Each telephone check-in session will last approximately 30-45 minutes and will include a brief review of the goals, a check in regarding the well-being of caregiver and PLWD and will address any questions or needs regarding post-discharge care navigation.

Caregiver study participant assessments will be conducted by telephone at baseline, at around 6 weeks (4-6 weeks depending on the availability of the caregiver), and at around 12 weeks (12-14 weeks depending on the availability of the caregiver) post-discharge. The GRA will also conduct chart reviews to gather additional patient outcome data. The primary outcomes of this pilot trial are acceptability, feasibility, and fidelity.

Interviews will be conducted with the CHW interventionist, palliative care team members, other primary care team members, information technology (IT) staff and/or other relevant staff at both study sites (DSMC and ASMCA) using in-depth interviews to explore acceptability and feasibility of the intervention. In addition, interviews will be conducted with key stakeholders and informants before and after the intervention is implemented. The goal of these interviews is to identify any additional challenges or priorities stakeholders experience during transitions of care that our intervention needs to consider. Stakeholders will include hospital staff from two sites (DSMC and ASMCA), content experts on dementia and caregiving (e.g., clinicians, service providers, scholars on this topic area), community organization providers for older adults and people living with dementia or their families, and formal or current dementia caregivers. Participants may be asked to participate in in-depth interviews multiple times, before the intervention is implemented, during the implementation period, and after the intervention has been implemented. Using a semi-structured interview (in person, phone, or zoom, whichever the participant prefers) which will take approximately 30-60 minutes.

To analyze the acceptability and feasibility of the protocol and barriers to recruitment and retention as well as systemwide implementation, analytic techniques for mixed methods study will be used such as content analyses and descriptive methods. All quantitative data analyses (e.g., descriptive, correlation,) will be conducted with SPSS v24 and R software. All qualitative interviews will be digitally-recorded and will be transcribed verbatim by a professional transcription service, and uploaded into Dedoose qualitative analysis software. A coding scheme and a codebook will be developed; codes will consist of externally-generated codes based on a predetermined conceptual framework, and internally-generated codes that emerge from the analysis with focus on codes reflecting potential difficulties with the intervention; opinions about the length and number of sessions; the delivery method; stakeholder priorities; implementation challenges and barriers; etc. Member checking will be ongoing from interview to interview. To corroborate findings and establish trustworthiness, an audit trail will be kept and co-investigators will be convened to provide critical feedback on the emerging codes. Data will be reviewed within and across coded texts in order to extract converging themes and reach consensus on principal themes.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized Patients:

1. Aged 50 or older
2. Has confirmed or suspected dementia or cognitive impairment (i.e., having memory concerns) ;
3. Has FAST score 4-6;
4. Admitted from home (not a long-term care facility)

Family Caregiver:

1. Aged 18 or older;
2. English or Spanish speaking;
3. Patient's relative, or partner who assists with medical care on a regular basis and who may or may not live in the same residence and who is not paid for their help; and
4. Legally authorized representative (LAR) for the patient if the patient is not able to consent for themselves in the study.

Staff Participants:

1. Aged 18 and older,
2. English speaking,
3. Employed full-time or part-time at or affiliated with either site, and
4. Involved directly or indirectly with patient care (i.e., administrative or non-clinical support staff) such as: nurses, physicians, physician assistants, care managers, social workers, chaplains, discharge planners, IT staff, administrative managers

Key Informants:

1. For hospital staff key informants, same eligibility criteria as above
2. For family caregivers (current or formal)

   1. Aged 18 or older;
   2. English or Spanish speaking;
   3. Currently or previously were caring for a relative with dementia

Content experts or community service providers:

1. Aged 18 or older;
2. English or Spanish speaking;
3. Have professional experience working with and/or have expertise about dementia care and caregiving or related areas (e.g., aging service providers, staff at Alzheimer's association, scholars in the area of aging, dementia, caregiving, or care transition)

Exclusion Criteria:

Hospitalized Patients:

1. Patients who do not meet eligibility criteria
2. Patients who are eligible for hospice

Caregivers:

1. Caregivers who do not meet the eligibility criteria

Staff participants:

1. Staff who do not meet the eligibility criteria
2. Staff who do not speak English

Key Informants:

1. Individuals who do not meet the eligibility criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Caregiver Acceptability | At post-discharge Week 12 follow up.
  Participants will be asked about acceptability using 7 items with Likert type scales which were developed by the research team to assess: (1) if the caregiver liked meetings with CHW (1=strongly dislike, 5=strongly like); (2) how much efforts the caregiver had to put in meeting with CHW (1=no effort at all, 5=huge effort); (3), if the CHW support was fair (1=very unfair, 5=very fair); (4) if the CHW support improved the patient experience (1=strongly disagree, 5=strongly agree); (5) if it was clear to the caregiver how the CHW support will improve the caregiver's ability to care for the patient (1=strongly disagree, 5=strongly agree); (6) how confident the caregiver was in participating meetings with the CHW (1=very unconfident, 5=very confident); and (7) overall rating of the acceptability of the intervention in support the caregiver (1=completely unacceptable, 5=completely acceptable).
Study Feasibility | Assessing feasibility begins with their enrollment (at Baseline) and ends with their final scheduled visit with the CHW (at Post-discharge Week 12 follow-up).
  Feasibility will be assessed by study enrollment rate (percentage of eligible persons enrolled in the study), and participant assessment completion rate (number of participants completing each study assessment at baseline, Post-discharge Week 6 and Post-discharge Week 12 follow-up). Consistent with other pilot intervention studies, 25% rate of enrollment, equal or higher than 70% completion rates for study assessments will be considered as evidence of feasibility.
Fidelity | CHW Initial Assessment Meeting (within the first week of enrollment), 1st CHW Follow-Up Meeting (within 4 weeks of the initial assessment meeting) and 2nd CHW Follow-Up Meeting (within 4 weeks of the 1st follow-up meeting)
  We will select approximately 20% of participants' interview recordings (at least one initial assessment and at least one follow-up CHW sessions), review and apply the fidelity checklist. The fidelity assessment was developed by the research team to evaluate CHW performance across key competencies using a structured scale. Nine items assess the CHW's skills and action including ability to accurately explain their role, convey a positive, non-judgmental attitude, active listening skills (e.g., reflection, validation, summarizing) and supportive responses to emotions are measured (scored 3 if consistent/always, 2 if inconsistent/sometimes, and 1 if absent/rarely). Four items assess presence of CHW following the crisis intervention model elements, e.g., facilitating the patient's immediate needs (scored 3 if present, 0 if absent). Assessment and follow-up form completeness is scored with 4 if 80% or higher, and 0 if less than 80%.
Intervention Feasibility | Baseline, Post-Discharge Week 6 Follow-up, Post-Discharge Week 12 Follow-up
  Feasibility will be assessed by intervention completion rate (number of participants completing the telephone sessions with the CHW ) Consistent with other pilot intervention studies, ≥70% completion rates for intervention session.

SECONDARY OUTCOMES:
PWLD quality of life | Post-Discharge Week 6 Follow-up, Post-Discharge Week 12 Follow-up
  PWLD quality of life is measured by Quality of Life in Alzheimer's Disease (QoL-AD) scale (Reference: Torisson G, Stavenow L, Minthon L, Londos E. Reliability, validity and clinical correlates of the Quality of Life in Alzheimer's Disease (QoL-AD) scale in medical inpatients. Health Qual Life Outcomes. 2016;14:90.)
PLWD 30- and 90- day hospital and ED readmissions | Post-Discharge Week 6 Follow-up, Post-Discharge Week 12 Follow-up
  PLWD's 30- and 90- day hospital and ED readmission rate will be assessed by asking the caregiver to report during the interview. They will be asked: how many times the PLWD was admitted to a hospital for any reason in the last 30 days and last 90 days and how many times the PLWD was admitted to an ER for any reason in the last 30 days and last 90 days.
Caregiver burden | Post-discharge Week 6 Follow-up, Post-discharge Week 12 Follow-up
  Caregiver burden will be measured by the Zarit Burden Short Interview (Reference: Michel Bédard, D. William Molloy, Larry Squire, Sacha Dubois, Judith A. Lever, Martin O'Donnell, The Zarit Burden Interview: A New Short Version and Screening Version, The Gerontologist, Volume 41, Issue 5, 1 October 2001, Pages 652-657, https://doi.org/10.1093/geront/41.5.652)
Caregiver well-being | Post-discharge Week 6 Follow-up and Post-discharge Week 12 Follow-up
  Caregiver well-being will be measured by COPE scale (Reference: Aguirre, A., Benge, J.F., Finger, A., Ambiee, J., Runnels, I., Hilsabeck, R. (2024) The Caregiver Outcomes of Psychotherapy Evaluation (COPE): Development of a Social Work Assessment Tool. Clinical Social Work Journal. https://doi.org/10.1007/s10615-024-00925-2)
Care transition quality | Post-discharge Week 6 Follow-up, Post-discharge Week 12 Follow-up
  Care transition quality will be measured by the Family Caregiver Activation in Transitions (FCAT) Tool (Reference: Coleman EA, Ground KL, Maul A. The Family Caregiver Activation in Transitions (FCAT) Tool: A New Measure of Family Caregiver Self-Efficacy. Jt Comm J Qual Patient Saf. 2015;41(11):502-507.)
Post-discharge compliance | Post-discharge Week 6 Follow-up, Post-discharge Week 12 Follow-up
  Post-discharge compliance will be measured by items adapted from Albrecht et al's discharge instruction comprehension measure about medications, follow-up appointments, diet, and exercise (Reference: Albrecht JS, Gruber-Baldini AL, Hirshon JM, et al. Hospital Discharge Instructions: Comprehension and Compliance Among Older Adults. J Gen Intern Med. 2014;29(11):1491-1498.)

CONTACTS AND LOCATIONS:
Overall Officials: Jung Kwak, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- Dell Seton Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All raw data accessibility will be limited to the PI, data manager, GRAs, and the statistician.
  Data will be shared under a two-tier distribution system. All data that can be de-identified will be shared. Data with specific confidentially risks, such as individual-level digital recordings will not be shared publicly because of the difficulty masking the identity of participants. Data with increased risk of reidentification will be shared under a data-use agreement that clearly establish use rules to facilitate respondent confidentiality.
  Even though the final dataset comprising of questionnaire will be stripped of identifiers prior to release for sharing, we believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics. These types of data will be only shared under a data sharing agreement: individual-level digital recordings, medical records review, and qualitative data from participants interviews (because of the difficulty masking).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start date: January 1, 2027; end date: December 31, 2029
Access Criteria: All raw data accessibility will be limited to the PI, data manager, GRAs, and the statistician. Data will be shared under a two-tier distribution system. All data that can be de-identified will be publicly shared. Data with increased risk of reidentification will be shared under a data-use agreement that clearly establish use rules to facilitate respondent confidentiality. We will make these data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. After review of the purpose of the data request to make sure it is consistent with the original project goals and verification that the request meets IRB approval, de-identified data may be shared with researchers.

REFERENCES:
- [Background] Kwak J, Kvale E, Mills S, Patel S. Co-designing a stage 1B feasibility study of inpatient palliative community health worker support. Innov Aging. 2023;7(suppl 1):337-338. https://doi.org/10.1093/geroni/igad104.1124
- [Derived] Kwak J, Jafari A, Salter A, Perry A, de Montfort Shepherd A, Jayasundera M, Stayer S, Brode M, Patel S, Kvale E. CEDART Study: protocol for a non-randomized feasibility study. Res Sq [Preprint]. 2025 May 13:rs.3.rs-6378596. doi: 10.21203/rs.3.rs-6378596/v1. PMID 40470215